CLINICAL TRIAL: NCT00878020
Title: Randomized, Double-Blind, Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BMS-830216 (Pro-Drug of BMS-819881) in Healthy Subjects
Brief Title: Safety Study to Evaluate BMS-830216 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB123-001
Record Dates: First submitted 2009-04-02; First posted 2009-04-08 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2009-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Active Comparator): BMS-830216 (10 mg)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Arm 2 (Active Comparator): BMS-830216 (30 mg)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Arm 3 (Active Comparator): BMS-830216 (100 mg)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Arm 4 (Active Comparator): BMS-830216 (300 mg)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Arm 5 (Active Comparator): BMS-830216 (600 mg)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Arm 6 (Active Comparator): BMS-830216 (1200 mg)
  Interventions: Drug: BMS-830216; Drug: Placebo

INTERVENTIONS:
Drug: BMS-830216 — Capsules, Oral, Single Dose, 1 day
  Arms: Arm 1; Arm 2; Arm 3; Arm 5; Arm 6
Drug: Placebo — Capsules, Oral, 0mg, Single Dose, 1 day
  Arms: Arm 1; Arm 2; Arm 3; Arm 5; Arm 6
Drug: BMS-830216 — Capsules, Oral, Single Dose on Day 1, Period 1 and Day 1, Period 2, 2 days
  Arms: Arm 4
Drug: Placebo — Capsules, Oral, 0mg, Single Dose, on Day 1, Period 1 and Day 1, Period 2, 2 days
  Arms: Arm 4

SUMMARY:
The purpose of this study is to evaluate the safety profile, tolerability, and pharmacokinetics of single oral doses from 10 mg up to 1200 mg of BMS-830216 (pro-drug of BMS-819881) in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects as determined by medical history, physical examination, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations will be eligible to participate in the study
* Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and men between ages of 18 to 45

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs), vital signs, electrocardiogram (ECG) and clinical laboratory test results | Within the 10 days after study drug administration

SECONDARY OUTCOMES:
Pharmacokinetic profile (drug absorption, distribution, metabolism and excretion process) determined by plasma concentration vs. time profile from a series of plasma samples up to 10 days post dose | Within the 10 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx